CLINICAL TRIAL: NCT04340882
Title: A Phase 2 Study of Docetaxel, Ramucirumab, and Pembrolizumab for Patients With Metastatic or Recurrent Non-Small Cell Lung Cancer Who Progressed on Platinum-Doublet and PD-1/PD-L1 Blockade
Brief Title: Phase 2 DoceRamPem for Patients With Metastatic or Recurrent NSCLC Who Progressed on Platinum-Doublet and PD-1/PD-L1 Blockade
Acronym: DoceRamPem
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Badi El Osta, MD, FACP, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000030; NCI-2020-01134 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); WINSHIP4950-20 (Other: Emory University); P30CA138292 (NIH)
Record Dates: First submitted 2020-04-07; First posted 2020-04-10 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Non-Small Lung Cell Cancer; Recurrent Non-Small Lung Cell Cancer; Stage IV Lung Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8
MeSH Terms: conditions — Lung Neoplasms | interventions — Docetaxel; pembrolizumab; Ramucirumab

STUDY DESIGN:
Intervention Model Description: Phase 2 with initial run-in safety
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (docetaxel, ramucirumab, pembrolizumab) (Experimental): Patients receive docetaxel IV over 60 minutes, ramucirumab IV over 60 minutes, and pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Docetaxel; Biological: Pembrolizumab; Biological: Ramucirumab

INTERVENTIONS:
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP56976; Taxotere; Taxotere Injection Concentrate
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Biological: Ramucirumab — Given IV
  Other Names: Anti-VEGFR-2 Fully Human Monoclonal Antibody IMC-1121B; Cyramza; IMC-1121B; LY3009806; Monoclonal Antibody HGS-ETR2

SUMMARY:
This phase 2 trial will evaluate the safety and efficacy of combining immunotherapy with a PD-1 checkpoint inhibitor (Pembrolizumab), an anti-VEGF receptor (Ramucirumab), and a taxane chemotherapy (Docetaxel) in treating patients with non-small cell lung cancer (NSCLC) who did not respond to FDA-approved treatments with platinum-based chemotherapy given concurrently or sequentially with anti-PD1/PD-L1 immunotherapy.

Pembrolizumab helps the body's immune system to attack cancer cells and hinder their ability to grow and spread. Ramucirumab blocks new blood vessel growth to reduce tumor growth. Docetaxel works mainly by stopping cancer cells from dividing. Ramucirumab combined with docetaxel is an FDA-approved therapy for NSCLC patients after progression on platinum-based chemotherapy. It has shown to improve efficacy compared to docetaxel alone in this setting. Pembrolizumab is an FDA-approved treatment for NSCLC and can be given alone or in combination with platinum-based chemotherapy.

Investigators hypothesize that the combination of docetaxel, ramucirumab, and pembrolizumab will be safe and more effective than the current standard of care treatments (docetaxel alone or in combination with ramucirumab) in patients with metastatic or recurrent NSCLC after progression on treatment with platinum-based chemotherapy and immunotherapy, given concurrently or sequentially.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the anti-tumor efficacy of the combination treatment using the 6-month progression free survival rate by Response Evaluation Criteria in Solid Tumors (RECIST 1.1).

SECONDARY OBJECTIVES:

I. To determine the safety profile and tolerability of docetaxel and ramucirumab in combination with pembrolizumab in patients who progressed on platinum-based chemotherapy and PD-1 or PD-L1 checkpoint inhibitor given sequentially or in combination.

II. To determine immune related adverse events of the combination docetaxel, ramucirumab, and pembrolizumab.

III. To assess the overall response rate (ORR) of the combination docetaxel, ramucirumab, and pembrolizumab.

IV. To assess the overall survival (OS) of the combination docetaxel, ramucirumab, and pembrolizumab.

EXPLORATORY OBJECTIVES:

I. To correlate treatment response with PD-L1 22C3 expression, STK11 and KRAS mutation status.

II. To correlate treatment response with the doublet tumor mutation burden (TMB) and PD-L1 22C3 expression.

III. To perform an immunophenotypic analysis of circulating immune cells by mass cytometry before and after treatment and end of treatment (EOT).

IV. To analyze the tumor infiltrating immune cells by mass cytometry coupled to blood mass cytometry, in paired biopsies before and at end of after treatment.

OUTLINE:

After premedication, patients will receive docetaxel intravenously (IV) over 60 minutes, ramucirumab IV over 60 minutes, then pembrolizumab IV over 30 minutes on day 1 of each 21-day cycle. The combination will be administered until confirmed disease progression defined as progression on 2 consecutive scans at least 4 weeks apart, occurrence of severe side effects, withdrawal of consent by the patient or if in the opinion of the treating physician continuing on the study treatment is not in the best interest of the patient.

The first six patients will be evaluated for safety data. If less than 2 patients experience dose limiting toxicity, enrollment on study will continue with the efficacy assessment of the combination.

Participants who experience confirmed disease progression or start a new anticancer therapy, will move into the Survival Follow-Up Phase and should be contacted by telephone every 12 weeks (+/- 3 weeks) for 2 years, then every 6 months for next 3 years, then annually until the subject's death or until the subject is lost to follow-up up to 10 years to assess for survival status until death, withdrawal of consent, or the end of the trial, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of non-small cell lung cancer
* Patients must have progressed on a platinum-based chemotherapy and any of the Food and Drug Administration (FDA)-approved PD-1 or PD-L1 immune checkpoint inhibitors, either given sequentially or in combination
* A male participant must agree to use a contraception during the treatment period plus an additional 120 days after the last dose of study treatment and refrain from donating sperm during this period
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

  * Not a woman of childbearing potential (WOCBP) OR
  * A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 120 days plus 30 days (a menstruation cycle) after the last dose of study treatment
* The participant (or legally acceptable representative if applicable) provides written informed consent for the trial
* Has measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Life expectancy > 12 weeks as determined by the investigator
* Absolute neutrophil count (ANC) ≥ 1500/uL (collected within 10 days prior to the start of study treatment)
* Platelets ≥ 100 000/uL (collected within 10 days prior to the start of study treatment)
* Hemoglobin ≥ 9.0 g/dL or ≥ 5.6 mmol/L (collected within 10 days prior to the start of study treatment)

  * Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks
* Creatinine ≤ 1.5 x upper limit of normal (ULN) OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) ≥ 30 mL/min for participant with creatinine levels > 1.5 x institutional ULN (collected within 10 days prior to the start of study treatment)

  * Creatinine clearance (CrCl) should be calculated per institutional standard
* Total bilirubin ≤ 1.5 x ULN OR direct bilirubin ≤ ULN for participants with total bilirubin levels > 1.5 x ULN (collected within 10 days prior to the start of study treatment)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) ≤ 2.5 x ULN (≤ 5 x ULN for participants with liver metastases) (collected within 10 days prior to the start of study treatment
* Palliative radiotherapy (to bone or soft tissue lesions) must be completed > 1 week prior to start of study drug (exception: palliative radiotherapy for pain may be used any time prior to first dose)
* Clinically significant toxic effect(s) of the most recent prior anti-cancer therapy must be grade 1 or resolved (except alopecia and sensory neuropathy); patients with grade 2 adrenal insufficiency related to prior anti-cancer therapy (defined as requiring medical intervention, such as concomitant steroids) or grade 2 hypothyroidism (defined as requiring hormone replacement therapy) may be enrolled provided that clinical symptoms are adequately controlled and the daily dose is 10 mg or less of prednisone or equivalent. If the patient received major surgery or radiation therapy of > 30 Gy, they must have recovered from the toxicity and/or complications from the intervention
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better

Exclusion Criteria:

* A WOCBP with a positive urine pregnancy test within 72 hours prior of the planned treatment on day 1 of each cycle. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Patients have prior exposure to docetaxel or ramucirumab
* Patients with proteinuria of ≥ 2+ on dipsticks or urine protein/creatinine ratio of > 1 g/24-hour
* Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks or 5 times the half-life time, whichever is shorter [could consider shorter interval for kinase inhibitors or other short half-life drugs] prior to allocation

  * Note: Participants must have recovered from all adverse events (AEs) due to previous therapies to grade ≤ 1 or baseline. Participants with grade ≤ 2 neuropathy may be eligible
  * Note: If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment
* Has received prior radiotherapy within 1 week of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤ 2 weeks of radiotherapy) to non-central nervous system (CNS) disease
* Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, bacillus Calmette-Guerin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist) are live attenuated vaccines and are not allowed
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment

  * Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug
* Patients with symptomatic brain metastasis (patients with treated brain metastasis without symptoms and not requiring steroid are allowed to participate)
* Has severe hypersensitivity (grade ≥ 3) to pembrolizumab and/or any of its excipients
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, significant cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients with significant cardiovascular disease (e.g., myocardial infarction, arterial thromboembolism, cerebrovascular thromboembolism) within 6 months prior to start of study therapy; angina requiring therapy; symptomatic peripheral vascular disease; New York Heart Association class 3 or 4 congestive heart failure; or uncontrolled grade ≥ 3 hypertension (diastolic blood pressure ≥ 100 mmHg or systolic blood pressure ≥ 160 mmHg) despite antihypertensive therapy
* Patients with any major hemorrhage or thromboembolic events within 3 months prior to start on this study
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis or established interstitial lung disease
* Patients who had prior history of immune-related adverse event (irAE) that required treatment with steroids and permanent immune checkpoint inhibitor (ICI) discontinuation per National Comprehensive Cancer Network (NCCN) guidelines
* Has an active infection requiring systemic therapy
* Has a known history of Human Immunodeficiency Virus (HIV). Note: no HIV testing is required unless mandated by local health authority
* Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-06-05 (Actual); Primary Completion 2026-09-02 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
6-month progression-free survival (PFS) rate | up to 6 months
  Will be determined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Will be reported and its 95% confidence intervals will be estimated using the Clopper-Pearson method. PFS rates of two patient groups stratified by binary biomarker (PD-L1 and KRAS status), respectively will be estimated with the Kaplan-Meier method and compared using the log-rank test, respectively. Cox proportional hazards models will be further used in the multivariable analyses to assess adjusted effect of PD-L1 and KRAS status on the patients' PFS after adjusting for other factors. Interaction terms between these factors will also be tested for statistical significance. The proportional hazards assumption will be evaluated graphically and analytically with regression diagnostics. Violations of the proportional hazards assumptions will be addressed by use of time-dependent covariates or extended Cox regression models.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 30 days after the last dose of study treatment
  Will be evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. Overall toxicity incidence as well as toxicity profiles will be explored and summarized. Frequency distributions, graphical techniques and other descriptive measures will form the basis of these analyses. Proportion of acute and late toxicity will be reported, and 95% confidence intervals will be estimated using the Clopper-Pearson method.
Overall response rate | Through study completion, an average of 1 year
  Will be determined per RECIST 1.1 and immune-modified Response Evaluation Criteria in Solid Tumors.
Overall survival (OS) | up to 10 years
  OS and rates of two patient groups stratified by binary biomarker (PD-L1 and KRAS status), respectively will be estimated with the Kaplan-Meier method and compared using the log-rank test, respectively. Cox proportional hazards models will be further used in the multivariable analyses to assess adjusted effect of PD-L1 and KRAS status on the patients' OS after adjusting for other factors. Interaction terms between these factors will also be tested for statistical significance. The proportional hazards assumption will be evaluated graphically and analytically with regression diagnostics. Violations of the proportional hazards assumptions will be addressed by use of time-dependent covariates or extended Cox regression models.

CONTACTS AND LOCATIONS:
Overall Officials: Badi El Osta, MD, FACP, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Grady Health System, Atlanta, Georgia
  - Winship Cancer Institute of Emory University, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No
Results of the trial and not individual patient data will be shared. The study protocol, consent, and investigator's brochure will be available. The statistical plan is incorporated into the protocol, along with inclusion and exclusion criteria.

REFERENCES:
- [Background] Osta BE, Carlisle J, Steuer C, Pakkala S, Leal T, Dhodapkar M, Liu Y, Chen Z, Owonikoko T, Ramalingam S. A Phase 2 Study of Docetaxel, Ramucirumab, and Pembrolizumab for Patients With Metastatic or Recurrent Non-Small-Cell Lung Cancer (NSCLC) who Progressed on Platinum-Doublet and PD-1/PD-L1 Blockade. Clin Lung Cancer. 2022 Nov;23(7):e400-e404. doi: 10.1016/j.cllc.2022.06.003. Epub 2022 Jun 22. PMID 35863963

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-03-07): https://cdn.clinicaltrials.gov/large-docs/82/NCT04340882/Prot_SAP_000.pdf
  • Informed Consent Form (2025-02-07): https://cdn.clinicaltrials.gov/large-docs/82/NCT04340882/ICF_001.pdf